CLINICAL TRIAL: NCT06187844
Title: Value of Inguinal Exploration in Cases of Impalpable Testis With Cord Structures Entering the Inguinal Canal
Brief Title: Value of Inguinal Exploration for Impalpable Testes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Omar Mohamed, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: expl impalpable testes
Record Dates: First submitted 2023-10-06; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Undescended Testis; Inguinal; Testicle
MeSH Terms: conditions — Cryptorchidism | interventions — Laparoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with impalpable tests (Experimental): For children with impalpable tests before and under anesthesia and by laparoscopy, cord structures could be seen entering the inguinal canal, inguinal exploration will be done.
  Interventions: Procedure: Inguinal exploration; Procedure: Laparoscopy

INTERVENTIONS:
Procedure: Inguinal exploration — Inguinal exploration will be done for all the included patients.
Procedure: Laparoscopy — All patients will have abdominal laparoscopy first to assess the location of the impalpable testis, the inguinal canal and the cord structures.

SUMMARY:
* To determine the percentage of children with impalpable testis who benefit from inguinal exploration after laparoscopic identification of cord structures entering the inguinal canal.
* To determine the factors predicting the presence of inguinal testis in the previously mentioned children.

DETAILED DESCRIPTION:
The undescended testis represents one of the most common disorders of childhood. The most useful classification of undescended testes is distinguishing palpable and non-palpable tests, and the location and presence of the tests decide clinical management. Approximately 80% of all undescended tests are palpable and the other 20% are impalpable. Among the 20% of non-palpable testes, 50-60% are intra-abdominal, canalicular, or peeping (right inside the internal inguinal ring). The remaining 20% are absent and 30% are atrophic or rudimentary.

Diagnostic laparoscopy is the most useful modality for assessing nonpalpable testicles. The four most important structures to identify at laparoscopy are the testis, the testicular vessels, the vase deferens, and the patency of the processus vaginalis. The possible anatomical findings include spermatic vessels entering the inguinal canal (40%), an intra-abdominal (40%) or peeping (10%) testis, or blind-ending spermatic vessels confirming vanishing testis (10%). It permits the identification of three surgical scenarios that will lead to different courses of action:

1. Blind-ending vessels, which indicate a vanishing intra-abdominal testis, and no further exploration is necessary (10%)
2. Testicular vessels and vas entering the inguinal canal through the internal inguinal ring (34%).Inguinal exploration may find a testicular nubbin either in the inguinal region or in the scrotum, which may or may not be removed; or a healthy, palpable, undescended testicle amenable to standard orchidopexy.
3. Peeping (11%) or intra-abdominal tests (37%), which will require either an open or a laparoscopic approach. Although Rozanski et al. reported the first case of intratubular germ cell neoplasia originating from a testicular remnant, the necessity of removing nubbins is controversial.

ELIGIBILITY:
Inclusion Criteria:

* Age 6m-12y
* Impalpable tests (unilateral or bilateral)
* Laparoscopy: cord structures entering the inguinal canal.

Exclusion Criteria:

* Patient refusing participation in the study.
* Any contraindication to laparoscopy
* laparoscopy: cord structures passing through an open inguinal canal through which the laparoscopy could be advanced and visualize the tests.
* Disorders of sexual differentiation.
* Children whose tests became palpable under anesthesia and those with a history of previous inguinal canal exploration (hydrocele or hernia repair) or orchidopexy.

Ages: 6 Months to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
. Percentage of positive inguinal exploration even by finding a testis or nubbin | Intraoperative
  To determine the percentage of children with impalpable testis who get benefit from inguinal exploration after laparoscopic identification of cord structures entering the inguinal canal.
  Inguinal exploration may find a testicular nubbin either in the inguinal region or, most commonly, in the scrotum, which will be excised and sent for histopathology; or a healthy, palpable, undescended testicle amenable to standard orchidopexy.

SECONDARY OUTCOMES:
Association between these different factors and the presence of inguinal testis in whom impalpable by lap | Preoperative
  We will investigate the following factors that may predict the presence of inguinal tests, thus supporting or avoiding inguinal exploration.
  1. History of inguinal or scrotal exploration
  2. history of cryptorchidism
  3. BMI (weight and height will be combined to report BMI in kg/m^2)
  4. size of the other testis in cm
  5. scrotal compartment development
  6. palpable scrotal nubbin

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdel Hamed Metwaly, Ass. prof, Principal Investigator — Assiut University

REFERENCES:
- [Background] Riedmiller H, Androulakakis P, Beurton D, Kocvara R, Gerharz E; European Association of Urology. EAU guidelines on paediatric urology. Eur Urol. 2001 Nov;40(5):589-99. doi: 10.1159/000049841. No abstract available. PMID 11752871
- [Background] Fratric I, Sarac D, Antic J, Dermanov M, Jokic R. Impalpable Testis: Evaluation of Diagnostic and Treatment Procedures and Our Treatment Protocol. Biomed Res Int. 2018 Jul 17;2018:3143412. doi: 10.1155/2018/3143412. eCollection 2018. PMID 30112376
- [Background] Van Savage JG. Avoidance of inguinal incision in laparoscopically confirmed vanishing testis syndrome. J Urol. 2001 Oct;166(4):1421-4. doi: 10.1097/00005392-200110000-00060. PMID 11547102
- [Background] Braga LH, Kim S, Farrokhyar F, Lorenzo AJ. Is there an optimal contralateral testicular cut-off size that predicts monorchism in boys with nonpalpable testicles? J Pediatr Urol. 2014 Aug;10(4):693-8. doi: 10.1016/j.jpurol.2014.05.011. Epub 2014 Jun 20. PMID 25008806
- [Background] Ueda N, Shiroyanagi Y, Suzuki H, Kim WJ, Yamazaki Y, Tanaka Y. The value of finding a closed internal ring on laparoscopy in unilateral nonpalpable testis. J Pediatr Surg. 2013 Mar;48(3):542-6. doi: 10.1016/j.jpedsurg.2012.09.032. PMID 23480909
- [Background] Rozanski TA, Wojno KJ, Bloom DA. The remnant orchiectomy. J Urol. 1996 Feb;155(2):712-3; discussion 714. PMID 8558712